CLINICAL TRIAL: NCT02817828
Title: A Multicenter, Open-label, Single-Arm Study to Evaluate the Contraceptive Efficacy and Safety of a Combined Oral Contraceptive Containing 15 mg Estetrol and 3 mg Drospirenone
Brief Title: E4 FREEDOM (Female Response Concerning Efficacy and Safety of Estetrol/Drospirenone as Oral Contraceptive in a Multicentric Study) - EU/Russia Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Estetra (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MIT-Es0001-C301
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Contraception
Keywords: Estetrol
MeSH Terms: interventions — Estetrol; drospirenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 15 mg E4/3 mg DRSP (Experimental): 15 mg E4/3 mg DRSP tablet
  Interventions: Drug: 15 mg E4/3 mg DRSP

INTERVENTIONS:
Drug: 15 mg E4/3 mg DRSP — 15 mg estetrol and 3 mg drospirenone tablets administered once daily for 13 consecutive cycles following a 24/4-day regimen, i.e. one 15 mg E4/3 mg DRSP active tablet per day for 24 consecutive days followed by one placebo tablet per day for 4 consecutive days.
  Other Names: 15 mg estetrol and 3 mg drospirenone

SUMMARY:
The objectives of this study are to evaluate the contraceptive efficacy, vaginal bleeding pattern (cycle control), and the general safety and acceptability of the 15 mg estetrol (E4)/3 mg drospirenone (DRSP) combination in healthy women aged 18 to 50 years.

ELIGIBILITY:
Inclusion Criteria:

* Heterosexually active female at risk for pregnancy and requesting contraception.
* Negative serum pregnancy test at subject enrollment.
* Willing to use the investigational product as the primary method of contraception for 13 consecutive cycles.
* Good physical and mental health on the basis of medical, surgical and gynecological history, physical examination, gynecological examination, clinical laboratory, and vital signs.
* Body mass index (BMI) below or equal to (≤) 35.0 kg/m2.
* Able to fulfill the requirements of the protocol and have indicated a willingness to participate in the study by providing written informed consent (IC).
* Willing and able to complete the diaries and questionnaires.

Exclusion Criteria:

* Known hypersensitivity to any of the investigational product ingredients.
* Smoking if ≥ 35 years old, at screening.
* Any condition associated with decrease fertility.
* Dyslipoproteinemia requiring active treatment with antilipidemic agent.
* Diabetes mellitus with vascular involvement (nephropathy, retinopathy, neuropathy, other) or diabetes mellitus of more than 20-year duration.
* Arterial hypertension.
* Any condition associated with an increased risk of venous thromboembolism and/or arterial thromboembolism.
* Any condition associated with abnormal uterine/vaginal bleeding.
* Abnormal Pap test based on current international recommendations.
* Presence of an undiagnosed breast mass.
* Current symptomatic gallbladder disease.
* History of COC related cholestasis.
* Presence or history of severe hepatic disease.
* Presence or history of pancreatitis if associated with hypertriglyceridemia.
* Porphyria.
* Presence or history of hepatocellular adenoma or malignant liver tumors.
* Renal impairment.
* Hyperkaliemia or presence of conditions that predispose to hyperkaliemia.
* Presence or history of hormone-related malignancy.
* History of non-hormone-related malignancy within 5 years before screening. Subjects with a non-melanoma skin cancer are allowed in the study.
* Use of drugs potentially triggering interactions with COCs.
* History of alcohol or drug abuse (including laxatives) within 12 months prior to screening.
* Any condition that could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the investigational product.
* Uncontrolled thyroid disorders.
* Participation in another investigational drug clinical study within 1 month (30 days) or have received an investigational drug within the last 3 months (90 days) prior to study entry. Subjects who participated in an oral contraceptive clinical study, using FDA/EU approved active ingredients, may be enrolled 2 months (60 days) after completing the preceding study.
* Sponsor, CRO or Investigator's site personnel directly affiliated with this study.
* Is judged by the Investigator to be unsuitable for any reason.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1577 (Actual)
Dates: Start 2016-06; Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Estetra, Study Director — Estetra
Locations (1):
- Hopital Saint-Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Creinin MD, Jensen JT, Chen MJ, Black A, Costescu D, Foidart JM. Combined Oral Contraceptive Adherence and Pregnancy Rates. Obstet Gynecol. 2023 May 1;141(5):989-994. doi: 10.1097/AOG.0000000000005155. Epub 2023 Apr 5. PMID 37023457

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1,577 participants aged 18-50 years were enrolled. Of those, 1,553 started the study treatment. Twenty-four participants did not start the treatment for the following reasons: consent withdrawn (8), unspecified reason (5), protocol deviation (3), pregnancy (4), lost to follow-up (3), and adverse event not related to bleeding (1).
Groups:
- 15 mg E4/3 mg DRSP: 15 mg E4/3 mg DRSP tablet
  15 mg E4/3 mg DRSP: 15 mg estetrol and 3 mg drospirenone tablets administered orally once daily for 13 consecutive cycles following a 24/4-day regimen, i.e. one 15 mg E4/3 mg DRSP active tablet per day for 24 consecutive days followed by one placebo tablet per day for 4 consecutive days.
Period: Overall Study
Arm/Group | 15 mg E4/3 mg DRSP
Started | 1553
Completed | 1218
Not Completed | 335
Not completed — Lost to Follow-up | 41
Not completed — Adverse event not related to bleeding | 104
Not completed — Adverse event related to bleeding | 53
Not completed — Protocol Violation | 11
Not completed — Pregnancy | 7
Not completed — Pregnancy wish | 15
Not completed — Withdrawal by Subject | 78
Not completed — Other | 26

BASELINE CHARACTERISTICS:
Population: All participants aged 18 to 50 years who received at least one dose of 15 mg E4/3 mg DRSP
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,553
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1,553
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (6.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1,553
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 1540
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 87
  Czechia | 335
  Finland | 181
  Germany | 141
  Hungary | 190
  Norway | 108
  Poland | 221
  Russia | 280
  Sweden | 10
Body mass index [Mean (Standard Deviation); unit: Kg/m^2] | 23.0 (3.469)

OUTCOME MEASURES:

1. Primary Outcome: The Number of On-treatment Pregnancies (With + 2-day Window) Per 100 Woman-years of Exposure (Pearl Index) in Subjects Aged 18 to 35 Years, Inclusive, at the Time of Screening
Description: On-treatment pregnancies are defined as pregnancies with an estimated date of conception within the in-treatment period i.e. Day 1 to 2 days after the last intake of investigational product (whether active or inactive tablet). The Pearl Index, defined as the number of pregnancies per 100 women-years of treatment was calculated as: Pearl Index = (1300*number of on-treatment pregnancies)/number of women 28-day equivalent cycles of treatment.Only at-risk cycles were included in the denominator of the Pearl Index calculation.
  At-risk-cycles were defined as cycles in which no other methods of birth control (including condoms) were used by the subject as confirmed in the subject diary and during which the subject confirmed that sexual intercourse had occurred.
Time Frame: Up to 12 months (13 cycles with 1 cycle = 28 days)
Population: Participants aged 18 to 35 years, inclusive, at screening with at least 1 cycle included in the denominator.
Measure: Number (95% Confidence Interval); unit: Pearl Index
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,313
Pearl Index | 0.47 [0.15 to 1.11]

2. Secondary Outcome: The Number of On-treatment Pregnancies (With 2-day Window) as Assessed by the Method Failure Pearl Index in Subjects Aged 18 to 35 Years, Inclusive, at the Time of Screening
Description: On-treatment pregnancies are defined as pregnancies with an estimated date of conception within the in-treatment period i.e. Day 1 to 2 days after the last intake of investigational product (whether active or inactive tablet). The Pearl Index, defined as the number of pregnancies per 100 women-years of treatment was calculated as: Pearl Index = (1300*number of on-treatment pregnancies)/number of women 28-day equivalent cycles of treatment. The method failure Pearl Index includes only those pregnancies that were classified as method failure and not the pregnancies due to user failure, i.e. incorrect intake of the contraceptive method. Only at-risk cycles were included in the denominator of the Pearl Index calculation. At-risk-cycles were defined as cycles in which no other methods of birth control (including condoms) were used by the subject as confirmed in the subject diary and during which the subject confirmed that sexual intercourse had occurred.
Time Frame: Up to 12 months (13 cycles with 1 cycle = 28 days)
Population: Participants aged 18 to 35 years, inclusive, at screening with at least 1 cycle included in the denominator.
Measure: Number (95% Confidence Interval); unit: Method failure Pearl Index
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,313
Method failure Pearl Index | 0.29 [0.06 to 0.83]

3. Secondary Outcome: The Number of On-treatment Pregnancies (With + 2-day Window) Per 100 Woman-years of Exposure (Pearl Index) in the Overall Study Population (18-50 Years)
Description: as for outcome 1
Time Frame: Up to 12 months (13 cycles with 1 cycle = 28 days)
Population: Participants aged 18 to 50 years, inclusive, at screening with at least 1 cycle included in the denominator.
Measure: Number (95% Confidence Interval); unit: Pearl Index
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,510
Pearl Index | 0.41 [0.13 to 0.96]

4. Secondary Outcome: The Number of On-Treatment Pregnancies as Assessed by the Method Failure Pearl Index in the Overall Study Population (18-50 Years)
Description: as for outcome 2
Time Frame: Up to 12 months (13 cycles with 1 cycle = 28 days)
Population: Participants aged 18 to 50 years, inclusive, at screening with at least 1 cycle included in the denominator.
Measure: Number (95% Confidence Interval); unit: Method Failure Pearl Index
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,510
Method Failure Pearl Index | 0.25 [0.05 to 0.72]

5. Secondary Outcome: Number of Subjects With Unscheduled Bleeding/Spotting
Description: Unscheduled bleeding/spotting is defined as any bleeding/spotting that occurs while taking active hormones that does not meet the criteria for scheduled bleeding.
Time Frame: Up to 11 months (12 cycles with 1 cycle = 28 days)
Population: Participants aged 18 to 50 years, inclusive, at screening, with evaluable cycle data for the bleeding analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,553
Participants
  Cycle 1: number analyzed (Participants) | 1,507
  Cycle 1 | 354
  Cycle 2: number analyzed (Participants) | 1,465
  Cycle 2 | 282
  Cycle 3: number analyzed (Participants) | 1,436
  Cycle 3 | 250
  Cycle 4: number analyzed (Participants) | 1,409
  Cycle 4 | 249
  Cycle 5: number analyzed (Participants) | 1,361
  Cycle 5 | 238
  Cycle 6: number analyzed (Participants) | 1,331
  Cycle 6 | 207
  Cycle 7: number analyzed (Participants) | 1,287
  Cycle 7 | 170
  Cycle 8: number analyzed (Participants) | 1,277
  Cycle 8 | 202
  Cycle 9: number analyzed (Participants) | 1,245
  Cycle 9 | 182
  Cycle 10: number analyzed (Participants) | 1,236
  Cycle 10 | 168
  Cycle 11: number analyzed (Participants) | 1,209
  Cycle 11 | 155
  Cycle 12: number analyzed (Participants) | 1,183
  Cycle 12 | 154

6. Secondary Outcome: Number of Unscheduled Bleeding Days Per Cycle
Description: Unscheduled bleeding is defined as any bleeding that occurs while taking active hormones that does not meet the criteria for scheduled bleeding and/or spotting.
Time Frame: Up to 11 months (12 cycles with 1 cycle = 28 days)
Population: Participants aged 18 to 50 years, inclusive, at screening, with evaluable cycle data for the bleeding analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,553
Days
  Cycle 1: number analyzed (Participants) | 1,507
  Cycle 1 | 0.2 (0.89)
  Cycle 2: number analyzed (Participants) | 1,465
  Cycle 2 | 0.1 (0.66)
  Cycle 3: number analyzed (Participants) | 1,436
  Cycle 3 | 0.1 (0.67)
  Cycle 4: number analyzed (Participants) | 1,409
  Cycle 4 | 0.2 (0.79)
  Cycle 5: number analyzed (Participants) | 1,361
  Cycle 5 | 0.1 (0.70)
  Cycle 6: number analyzed (Participants) | 1,331
  Cycle 6 | 0.1 (0.80)
  Cycle 7: number analyzed (Participants) | 1,287
  Cycle 7 | 0.1 (0.68)
  Cycle 8: number analyzed (Participants) | 1,277
  Cycle 8 | 0.1 (0.72)
  Cycle 9: number analyzed (Participants) | 1,245
  Cycle 9 | 0.1 (0.70)
  Cycle 10: number analyzed (Participants) | 1,236
  Cycle 10 | 0.1 (0.61)
  Cycle 11: number analyzed (Participants) | 1,209
  Cycle 11 | 0.1 (0.72)
  Cycle 12: number analyzed (Participants) | 1,183
  Cycle 12 | 0.1 (0.68)

7. Secondary Outcome: Number of Unscheduled Spotting Days Per Cycle
Description: Unscheduled spotting is defined as any spotting that occurs while taking active hormones that does not meet the criteria for scheduled bleeding and/or spotting.
Time Frame: Up to 11 months (12 cycles with 1 cycle = 28 days)
Population: Participants aged 18 to 50 years, inclusive, at screening, with evaluable cycle data for the bleeding analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,553
Days
  Cycle 1: number analyzed (Participants) | 1,507
  Cycle 1 | 0.8 (1.99)
  Cycle 2: number analyzed (Participants) | 1,465
  Cycle 2 | 0.5 (1.50)
  Cycle 3: number analyzed (Participants) | 1,436
  Cycle 3 | 0.5 (1.46)
  Cycle 4: number analyzed (Participants) | 1,409
  Cycle 4 | 0.5 (1.55)
  Cycle 5: number analyzed (Participants) | 1,361
  Cycle 5 | 0.5 (1.35)
  Cycle 6: number analyzed (Participants) | 1,331
  Cycle 6 | 0.4 (1.24)
  Cycle 7: number analyzed (Participants) | 1,287
  Cycle 7 | 0.4 (1.17)
  Cycle 8: number analyzed (Participants) | 1,277
  Cycle 8 | 0.4 (1.19)
  Cycle 9: number analyzed (Participants) | 1,245
  Cycle 9 | 0.4 (0.13)
  Cycle 10: number analyzed (Participants) | 1,236
  Cycle 10 | 0.4 (1.25)
  Cycle 11: number analyzed (Participants) | 1,209
  Cycle 11 | 0.3 (1.18)
  Cycle 12: number analyzed (Participants) | 1,183
  Cycle 12 | 0.4 (1.23)

8. Secondary Outcome: Number of Subjects With Absence of Scheduled Bleeding and/or Spotting
Description: Scheduled bleeding/spotting is defined as any bleeding/spotting that occurs during the hormone-free interval (i.e. Days 25 - 28) and continues through Days 1-3 of the subsequent active cycle.
Time Frame: Up to 11 months (12 cycles with 1 cycle = 28 days)
Population: Participants aged 18 to 50 years, inclusive, at screening, with evaluable cycle data for the bleeding analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,553
Participants
  Cycle 1: number analyzed (Participants) | 1,507
  Cycle 1 | 84
  Cycle 2: number analyzed (Participants) | 1,465
  Cycle 2 | 90
  Cycle 3: number analyzed (Participants) | 1,436
  Cycle 3 | 105
  Cycle 4: number analyzed (Participants) | 1,409
  Cycle 4 | 83
  Cycle 5: number analyzed (Participants) | 1,361
  Cycle 5 | 91
  Cycle 6: number analyzed (Participants) | 1,331
  Cycle 6 | 91
  Cycle 7: number analyzed (Participants) | 1,287
  Cycle 7 | 90
  Cycle 8: number analyzed (Participants) | 1,277
  Cycle 8 | 103
  Cycle 9: number analyzed (Participants) | 1,245
  Cycle 9 | 92
  Cycle 10: number analyzed (Participants) | 1,236
  Cycle 10 | 89
  Cycle 11: number analyzed (Participants) | 1,209
  Cycle 11 | 80
  Cycle 12: number analyzed (Participants) | 1,183
  Cycle 12 | 94

9. Secondary Outcome: Number of Scheduled Bleeding and/or Spotting Days Per Cycle
Description: Scheduled bleeding and /or spotting is defined as any bleeding and/or spotting that occurs during the hormone-free interval (i.e. Days 25 - 28) and continues through Days 1-3 of the subsequent active cycle.
Time Frame: Up to 11 months (12 cycles with 1 cycle = 28 days)
Population: Participants aged 18 to 50 years, inclusive, at screening, with evaluable cycle data for the bleeding analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,553
Days
  Cycle 1: number analyzed (Participants) | 1,507
  Cycle 1 | 6.1 (4.95)
  Cycle 2: number analyzed (Participants) | 1,465
  Cycle 2 | 5.3 (3.62)
  Cycle 3: number analyzed (Participants) | 1,436
  Cycle 3 | 5.2 (3.99)
  Cycle 4: number analyzed (Participants) | 1,409
  Cycle 4 | 5.0 (3.14)
  Cycle 5: number analyzed (Participants) | 1,361
  Cycle 5 | 4.9 (3.43)
  Cycle 6: number analyzed (Participants) | 1,331
  Cycle 6 | 4.9 (3.34)
  Cycle 7: number analyzed (Participants) | 1,287
  Cycle 7 | 4.7 (2.80)
  Cycle 8: number analyzed (Participants) | 1,277
  Cycle 8 | 4.8 (3.85)
  Cycle 9: number analyzed (Participants) | 1,245
  Cycle 9 | 4.7 (2.87)
  Cycle 10: number analyzed (Participants) | 1,236
  Cycle 10 | 4.6 (2.69)
  Cycle 11: number analyzed (Participants) | 1,209
  Cycle 11 | 4.7 (3.16)
  Cycle 12: number analyzed (Participants) | 1,183
  Cycle 12 | 4.6 (2.97)

10. Secondary Outcome: Number of Subjects With Abnormal Vital Signs
Description: Vital signs included sitting systolic and diastolic blood pressures, and heart rate.
Time Frame: From screening to end of treatment (12 months)
Population: Participants aged 18 to 50 years, inclusive, at screening, who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,553
Participants | 15

11. Secondary Outcome: Number of Subjects With Abnormal Laboratory Assessment Results
Description: Laboratory assessment included blood hematology, biochemistry, and lipids
Time Frame: From screening to end of treatment (12 months)
Population: Participants aged 18 to 50 years, inclusive, at screening, who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,553
Participants | 55

12. Secondary Outcome: Number of Subjects With Abnormal Physical Examination Results
Description: Physical examinations included an evaluation of body as a whole, skin, head, eyes, ears, nose, and throat, neck, cardiovascular, respiratory, musculoskeletal, neurologic, lymphatic/thyroid, abdomen.
  When reporting the results of the physical examination, the use of the "Abnormal" category was reserved for findings that were considered clinically significant, in the opinion of the Investigator; the "Normal" category included "Abnormal" results that were not clinically significant, as well as no findings.
Time Frame: From screening to end of treatment (12 months)
Population: Participants aged 18 to 50 years, inclusive, at screening, who received at least one dose of investigational product with baseline and end of treatment (EOT) results.
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,553
Participants
  Body as a whole - Baseline: Normal | 1548
  Body as a whole - Baseline: Abnormal | 5
  Body as a whole - Baseline: Not done | 0
  Body as a whole - EOT: number analyzed (Participants) | 1,498
  Body as a whole - EOT: Normal | 1493
  Body as a whole - EOT: Abnormal | 5
  Body as a whole - EOT: Not done | 0
  Skin - Baseline: Normal | 1537
  Skin - Baseline: Abnormal | 16
  Skin - Baseline: Not done | 0
  Skin - EOT: number analyzed (Participants) | 1,498
  Skin - EOT: Normal | 1,476
  Skin - EOT: Abnormal | 22
  Skin - EOT: Not done | 0
  Head, Eyes, Ears, Nose and Throat - Baseline: Normal | 1,543
  Head, Eyes, Ears, Nose and Throat - Baseline: Abnormal | 10
  Head, Eyes, Ears, Nose and Throat - Baseline: Not done | 0
  Head, Eyes, Ears, Nose and Throat - EOT: number analyzed (Participants) | 1,498
  Head, Eyes, Ears, Nose and Throat - EOT: Normal | 1,492
  Head, Eyes, Ears, Nose and Throat - EOT: Abnormal | 3
  Head, Eyes, Ears, Nose and Throat - EOT: Not done | 3
  Neck - Baseline: Normal | 1,552
  Neck - Baseline: Abnormal | 1
  Neck - Baseline: Not done | 0
  Neck - EOT: number analyzed (Participants) | 1,498
  Neck - EOT: Normal | 1,495
  Neck - EOT: Abnormal | 1
  Neck - EOT: Not done | 2
  Cardiovascular - Baseline: Normal | 1,553
  Cardiovascular - Baseline: Abnormal | 0
  Cardiovascular - Baseline: Not done | 0
  Cardiovascular - EOT: number analyzed (Participants) | 1,498
  Cardiovascular - EOT: Normal | 1,496
  Cardiovascular - EOT: Abnormal | 1
  Cardiovascular - EOT: Not done | 1
  Respiratory - Baseline: Normal | 1,551
  Respiratory - Baseline: Abnormal | 2
  Respiratory - Baseline: Not done | 0
  Respiratory - EOT: number analyzed (Participants) | 1,498
  Respiratory - EOT: Normal | 1,496
  Respiratory - EOT: Abnormal | 1
  Respiratory - EOT: Not done | 1
  Musculoskeletal - Baseline: Normal | 1,553
  Musculoskeletal - Baseline: Abnormal | 0
  Musculoskeletal - Baseline: Not done | 0
  Musculoskeletal - EOT: number analyzed (Participants) | 1,498
  Musculoskeletal - EOT: Normal | 1,495
  Musculoskeletal - EOT: Abnormal | 1
  Musculoskeletal - EOT: Not done | 2
  Neurologic - Baseline: Normal | 1,553
  Neurologic - Baseline: Abnormal | 0
  Neurologic - Baseline: Not done | 0
  Neurologic - EOT: number analyzed (Participants) | 1,498
  Neurologic - EOT: Normal | 1,494
  Neurologic - EOT: Abnormal | 2
  Neurologic - EOT: Not done | 2
  Lymphatic/Thyroid - Baseline: Normal | 1,549
  Lymphatic/Thyroid - Baseline: Abnormal | 2
  Lymphatic/Thyroid - Baseline: Not done | 2
  Lymphatic/Thyroid - EOT: number analyzed (Participants) | 1,498
  Lymphatic/Thyroid - EOT: Normal | 1,494
  Lymphatic/Thyroid - EOT: Abnormal | 1
  Lymphatic/Thyroid - EOT: Not done | 3
  Abdomen - Baseline: Normal | 1,553
  Abdomen - Baseline: Abnormal | 0
  Abdomen - Baseline: Not done | 0
  Abdomen - EOT: number analyzed (Participants) | 1,498
  Abdomen - EOT: Normal | 1,496
  Abdomen - EOT: Abnormal | 1
  Abdomen - EOT: Not done | 1

13. Secondary Outcome: Number of Subjects With Abnormal Gynecological Examination Results
Description: Gynecological examinations included breast examination (performed by palpation) and assessment of the adnexa, cervix, uterus, vagina, and external genitalia.
  When reporting the results, the use of the "Abnormal" category was reserved for findings that were considered clinically significant, in the opinion of the Investigator; the "Normal" category included "Abnormal" results that were not clinically significant, as well as no findings.
Time Frame: From screening to end of treatment (12 months)
Population: Participants aged 18 to 50 years, inclusive, at screening, who received at least one dose of investigational product with baseline and end of treatment (EOT) gynecological results.
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 1,553
Participants
  Breast - Baseline: Normal | 1,545
  Breast - Baseline: Abnormal | 8
  Breast - Baseline: Not done | 0
  Breast - EOT: number analyzed (Participants) | 1,499
  Breast - EOT: Normal | 1,485
  Breast - EOT: Abnormal | 13
  Breast - EOT: Not done | 1
  Adnexa - Baseline: Normal | 1,549
  Adnexa - Baseline: Abnormal | 4
  Adnexa - Baseline: Not done | 0
  Adnexa - EOT: number analyzed (Participants) | 1,499
  Adnexa - EOT: Normal | 1,496
  Adnexa - EOT: Abnormal | 2
  Adnexa - EOT: Not done | 1
  Cervix - Baseline: Normal | 1,532
  Cervix - Baseline: Abnormal | 21
  Cervix - Baseline: Not done | 0
  Cervix - EOT: number analyzed (Participants) | 1,499
  Cervix - EOT: Normal | 1,485
  Cervix - EOT: Abnormal | 13
  Cervix - EOT: Not done | 1
  Uterus - Baseline: Normal | 1,542
  Uterus - Baseline: Abnormal | 11
  Uterus - Baseline: Not done | 0
  Uterus - EOT: number analyzed (Participants) | 1,499
  Uterus - EOT: Normal | 1,492
  Uterus - EOT: Abnormal | 6
  Uterus - EOT: Not done | 1
  Vagina - Baseline: Normal | 1,545
  Vagina - Baseline: Abnormal | 8
  Vagina - Baseline: Not done | 0
  Vagina - EOT: number analyzed (Participants) | 1,499
  Vagina - EOT: Normal | 1,489
  Vagina - EOT: Abnormal | 8
  Vagina - EOT: Not done | 2
  External genitalia - Baseline: Normal | 1,552
  External genitalia - Baseline: Abnormal | 1
  External genitalia - Baseline: Not done | 0
  External genitalia - EOT: number analyzed (Participants) | 1,499
  External genitalia - EOT: Normal | 1,497
  External genitalia - EOT: Abnormal | 1
  External genitalia - EOT: Not done | 1

14. Secondary Outcome: Endometrial Biopsy Histology at Screening and End of Treatment
Description: Endometrial biopsies was obtained from a subset of subjects included in the endometrial safety substudy at the screening visit and at the end of treatment visit if the subject has completed at least 10 cycles.
Time Frame: Baseline and end of treatment (up to 13 cycles with 1 cycle = 28 days)
Population: Participants aged 18 to 50 years, inclusive, at screening with an evaluable endometrial biopsies both at screening and end of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | 15 mg E4/3 mg DRSP
Number analyzed (Participants) | 108
Participants
  Baseline: No tissue | 0
  Baseline: Tissue insufficient for diagnosis | 1
  Baseline: Benign histology:Atrophic | 2
  Baseline: Benign histology: Inactive | 7
  Baseline: Benign histology:Proliferative | 76
  Baseline: Secretory | 22
  Baseline: Menstrual type | 0
  Baseline: Simple hyperplasia without atypia | 0
  Baseline: Complex hyperplasia without atypia | 0
  Baseline: Pre-malignant/Malignant histology | 0
  End of Treatment: No tissue | 0
  End of Treatment: Tissue insufficient for diagnosis | 9
  End of Treatment: Benign histology:Atrophic | 11
  End of Treatment: Benign histology: Inactive | 61
  End of Treatment: Benign histology:Proliferative | 22
  End of Treatment: Secretory | 5
  End of Treatment: Menstrual type | 0
  End of Treatment: Simple hyperplasia without atypia | 0
  End of Treatment: Complex hyperplasia without atypia | 0
  End of Treatment: Pre-malignant/Malignant histology | 0

15. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) Results at Baseline and End of Treatment - Percentage Maximum (Sum of First 14 Items)
Description: The Q-LES-Q-SF is a self-report measure designed to assess the degree of enjoyment and satisfaction in daily functioning. Participants were asked to rate 16 different items on a 5-point scale where score 1 = very poor and score 5 = very good.
  A raw total score is calculated by summing the first 14 items and ranges from 14 to 70 with a higher scores indicating higher life enjoyment and satisfaction. The raw total score is then transformed into a percentage maximum score using the following formula: (raw total score-minimum score)/(maximum possible raw score-minimum score).
  In addition, the last two items (15 and 16) are two global items that are scored individually. These items rate "satisfaction with medicine" and "overall life satisfaction over the past week".
Time Frame: Baseline and Cycle 13 (1 cycle = 28 days)
Population: Participants aged 18 to 50 years, inclusive, at screening with baseline and end of treatment Q-LES-Q-SF results.
Measure: Mean (Standard Deviation); unit: Percentage maximum score on a scale
Groups:
- 15 mg E4/3 mg DRSP - Baseline Results; 15 mg E4/3 mg DRSP - End of Treatment Results: 15 mg E4/3 mg DRSP tablet
  15 mg E4/3 mg DRSP: 15 mg estetrol and 3 mg drospirenone tablets administered orally once daily for 13 consecutive cycles following a 24/4-day regimen, i.e. one 15 mg E4/3 mg DRSP active tablet per day for 24 consecutive days followed by one placebo tablet per day for 4 consecutive days.
Arm/Group | 15 mg E4/3 mg DRSP - Baseline Results | 15 mg E4/3 mg DRSP - End of Treatment Results
Number analyzed (Participants) | 1,379 | 1,406
Percentage maximum score on a scale | 73.4 (12.77) | 73.8 (12.82)

16. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) Results at Baseline and End of Treatment - Satisfaction With Medicine and Overall Life Satisfaction Over the Past Week
Description: as for outcome 15
Time Frame: Baseline and Cycle 13 (1 cycle = 28 days)
Population: Participants aged 18 to 50 years, inclusive, at screening with baseline and end of treatment Q-LES-Q-SF results.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 15 mg E4/3 mg DRSP - Baseline Results | 15 mg E4/3 mg DRSP - End of Treatment Results
Number analyzed (Participants) | 1,379 | 1,406
Units on a scale
  Satisfaction with medicine | 4.0 (0.78) | 4.0 (0.77)
  Overall life statisfaction over the past week | 4.0 (0.68) | 4.0 (0.70)

17. Secondary Outcome: Change From Baseline to End of Treatment in the Score of the Menstrual Distress Questionnaire (MDQ)
Description: The MDQ is a standard method for measuring cyclical perimenstrual symptoms. The participants rated common symptoms and feelings associated with menstruation using the following scale: 0 (no experience of symptom), 1 (present, mild), 2 (present, moderate), 3 (present, strong),and 4 (present, severe) observed during pre-menstrual (4 days before menstruation), menstrual (most recent flow) and intermenstrual (remainder of the cycle) phases.
  Reported values are values at Cycle 13 minus values at Baseline. An overall positive change from baseline represents an increase in symptom or feeling severity.
Time Frame: Baseline and Cycle 13 (1 cycle = 28 days)
Population: Participants aged 18 to 50 years, inclusive, at screening with both baseline and end of treatment MDQ results.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 15 mg E4/3 mg DRSP Tablet - Menstrual Phase; 15 mg E4/3 mg DRSP Tablet - Premenstrual Phase; 15 mg E4/3 mg DRSP Tablet - Intermenstrual Phase: 15 mg E4/3 mg DRSP tablet
  15 mg E4/3 mg DRSP: 15 mg estetrol and 3 mg drospirenone tablets administered orally once daily for 13 consecutive cycles following a 24/4-day regimen, i.e. one 15 mg E4/3 mg DRSP active tablet per day for 24 consecutive days followed by one placebo tablet per day for 4 consecutive days.
Arm/Group | 15 mg E4/3 mg DRSP Tablet - Menstrual Phase | 15 mg E4/3 mg DRSP Tablet - Premenstrual Phase | 15 mg E4/3 mg DRSP Tablet - Intermenstrual Phase
Number analyzed (Participants) | 1,553 | 1,553 | 1,553
units on a scale
  Pain: number analyzed (Participants) | 1,392 | 1,393 | 1,396
  Pain | -0.4 (3.6) | -0.1 (2.96) | -0.1 (2.67)
  Water retention: number analyzed (Participants) | 1,392 | 1,394 | 1,395
  Water retention | -0.1 (2.61) | -0.1 (2.57) | 0.0 (2.09)
  Autonomic reactions: number analyzed (Participants) | 1,392 | 1,393 | 1,396
  Autonomic reactions | -0.1 (1.42) | -0.0 (1.30) | -0.0 (1.22)
  Negative affect: number analyzed (Participants) | 1,392 | 1,393 | 1,395
  Negative affect | -0.4 (4.90) | -0.3 (4.70) | -0.1 (3.93)
  Impaired concentration: number analyzed (Participants) | 1,392 | 1,393 | 1,395
  Impaired concentration | 0.0 (2.67) | -0.0 (2.55) | 0.0 (2.23)
  Behaviour change: number analyzed (Participants) | 1,392 | 1,394 | 1,395
  Behaviour change | -0.1 (2.86) | -0.1 (2.55) | -0.0 (1.99)
  Arousal: number analyzed (Participants) | 1,392 | 1,393 | 1,395
  Arousal | -0.3 (3.46) | -0.3 (3.62) | -0.3 (3.91)
  Control: number analyzed (Participants) | 1,392 | 1,393 | 1,396
  Control | 0.0 (1.52) | 0.0 (1.57) | 0.0 (1.63)

ADVERSE EVENTS:
Time Frame: From screening to end of treatment (13 months)
Arm/Group | 15 mg E4/3 mg DRSP
All-Cause Mortality (participants affected / at risk) | 0/1553
Serious Adverse Events (participants affected / at risk) | 13/1553
Other Adverse Events (participants affected / at risk) | 784/1553
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg E4/3 mg DRSP (N=1553)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Migraine without aura (Nervous system disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2)
Abscess limb (Infections and infestations) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg E4/3 mg DRSP (N=1553)
Weight increased (Investigations) | 36 (36)
Low density lipoprotein increased (Investigations) | 18 (19)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 (16)
Dizziness (Nervous system disorders) | 19 (24)
Headache (Nervous system disorders) | 120 (171)
Mood altered (Nervous system disorders) | 19 (19)
Libido decreased (Nervous system disorders) | 38 (43)
Irritability (Nervous system disorders) | 18 (18)
Mood swings (Nervous system disorders) | 18 (18)
Abdominal pain (Gastrointestinal disorders) | 36 (48)
Diarrhoea (Gastrointestinal disorders) | 25 (45)
Vomiting (Gastrointestinal disorders) | 27 (49)
Nausea (Gastrointestinal disorders) | 20 (25)
Vaginal haemorrhage (Reproductive system and breast disorders) | 74 (151)
Dysmenorrhoea (Reproductive system and breast disorders) | 47 (74)
Metrorrhagia (Reproductive system and breast disorders) | 85 (156)
Breast pain (Reproductive system and breast disorders) | 42 (51)
Vaginal discharge (Reproductive system and breast disorders) | 16 (19)
Acne (Skin and subcutaneous tissue disorders) | 65 (69)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (20)
Tonsilitis (Infections and infestations) | 29 (31)
Vaginal infection (Infections and infestations) | 29 (33)
Influenza (Infections and infestations) | 28 (30)
Urinary tract infection (Infections and infestations) | 30 (35)
Vulvovaginal mycotic infection (Infections and infestations) | 17 (22)
Bronchitis (Infections and infestations) | 15 (16)
Sinusitis (Infections and infestations) | 17 (19)
Respiratory tract infection (Infections and infestations) | 18 (19)
Cystitis (Infections and infestations) | 24 (29)
Vulvovaginal candidiasis (Infections and infestations) | 20 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT02817828/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT02817828/SAP_001.pdf